CLINICAL TRIAL: NCT02893306
Title: Phase 2 Study of Intravenous Administration of Allogeneic Mesenchymal Stem Cells in Patients With Type 1 Diabetes Mellitus.
Brief Title: MSC Administration for the Management of Type 1 Diabetic Patients
Acronym: DMT1-MSC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad del Desarrollo (Other)
Collaborators: Clinica Alemana de Santiago (Other)
Responsible Party: Principal Investigator, Paulette Conget, Dr, Universidad del Desarrollo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMT1-MSC
Record Dates: First submitted 2016-08-27; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type1 Diabetes Mellitus; Multipotent stromal cell; Mesenchymal stem cell; Insulin; Pancreatic reserve; Disease progression
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DMT1+MSCs (Experimental): type 1 diabetic patients receiving a single dose of allogeneic ex vivo expanded mesenchymal stem cells
  Interventions: Biological: MSCs

INTERVENTIONS:
Biological: MSCs — origin: bone marrow of healthy donor; manipulation: ex vivo expanded; via: intravenous; vehicle: 5% human recombinant albumin in physiological serum; dose: 2-3 millions/Kg; dosage: single
  Other Names: mesenchymal stem cells

SUMMARY:
The purpose of this study is to evaluate whether the administration of multipotent stromal cell also referred as to mesenchymal stem cells (MSCs), modified Type 1 Diabetes progression.

DETAILED DESCRIPTION:
Aim: to evaluate whether a single intravenous administration of allogeneic bone marrow-derived multipotent stromal cell also referred as to mesenchymal stem cells (MSCs), modified endogenous insulin secretion capacity and exogenous insulin requirement in patients with Type 1 Diabetes Mellitus.

Participants: 10, females or males, 18 years or older, diagnosed with Type 1 Diabetes Mellitus at most 1 year before enrollment, under exogenous insulin treatment, with pancreatic reserve of insulin.

Intervention: intravenous administration of a single dose (2-3 millions/Kg) of allogeneic MSCs.

Follow up: before and 1, 6, 24 months after MSC administration.

ELIGIBILITY:
Inclusion Criteria:

* differential diagnosis of Type 1 Diabetes
* diagnosed performed at most 1 year before enrollment
* pancreatic reserve of insulin higher than 0.8 nmol/L/h
* good general health status
* informed consent of patient
* consent of treating physician
* proved psychiatric competence to be enrolled in a clinical study

Exclusion Criteria:

* pregnancy
* significant comorbidities
* HIV, HBV, HCV, HTLV-1, HLTV-2 or VDRL positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Changes in insulin pancreatic reserve | pre- and 1, 6, 24 months post-intervention
  Levels of insulin secreted after the acute ingestion of a protein rich liquid diet

SECONDARY OUTCOMES:
Changes in insulin requirement | pre- and up to 24 months post-intervention
  Daily dose of self-administered insulin

OTHER OUTCOMES:
Number of patients with grade 3 through grade 5 adverse events (CTCAE v3.0) | up to 24 months post-intervention
  Review of patient clinical records
Number of patients with grade 3 through grade 5 adverse events (CTCAE v3.0) | up to 24 months post-intervention
  Regular communication with patient and his/her physician in order to be informed of eventual complications

CONTACTS AND LOCATIONS:
Overall Officials: Paulette Conget, PhD, Principal Investigator — Universidad del Desarrollo; Claudio Mizon, MD, Principal Investigator — Clinica Alemana de Santiago
Locations (1):
- Clinica Alemana de Santiago, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Yes
Data will be publish in a peer review journal

REFERENCES:
- [Background] Ezquer F, Ezquer M, Contador D, Ricca M, Simon V, Conget P. The antidiabetic effect of mesenchymal stem cells is unrelated to their transdifferentiation potential but to their capability to restore Th1/Th2 balance and to modify the pancreatic microenvironment. Stem Cells. 2012 Aug;30(8):1664-74. doi: 10.1002/stem.1132. PMID 22644660
- [Background] Ezquer F, Ezquer M, Simon V, Conget P. The antidiabetic effect of MSCs is not impaired by insulin prophylaxis and is not improved by a second dose of cells. PLoS One. 2011 Jan 27;6(1):e16566. doi: 10.1371/journal.pone.0016566. PMID 21304603
- [Background] Ezquer FE, Ezquer ME, Parrau DB, Carpio D, Yanez AJ, Conget PA. Systemic administration of multipotent mesenchymal stromal cells reverts hyperglycemia and prevents nephropathy in type 1 diabetic mice. Biol Blood Marrow Transplant. 2008 Jun;14(6):631-40. doi: 10.1016/j.bbmt.2008.01.006. Epub 2008 Apr 14. PMID 18489988